CLINICAL TRIAL: NCT04909801
Title: A Randomized, Head-to-head, Single-blind Study to Compare the Response to Treatment With Subcutaneous Abatacept vs Adalimumab, on Background Methotrexate, in Adults With Early, Seropositive Rheumatoid Arthritis Who Have "Shared Epitope" HLA Class II Risk Alleles and Have an Inadequate Response to Methotrexate
Brief Title: A Study to Compare the Response to Treatment With Abatacept vs Adalimumab, on Background Methotrexate, in Adults With Early, Seropositive, and Shared Epitope-positive Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM101-863; 2020-000350-96 (EudraCT Number); U1111-1247-1367 (Registry Identifier: WHO)
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Abatacept; Adalimumab; BMS-188667; Humira®; Methotrexate; Orencia®; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Abatacept + Methotrexate (Experimental)
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Arm 2: (Adalimumab + Methotrexate) followed by (Abatacept + Methotrexate) (Experimental)
  Interventions: Drug: Abatacept; Drug: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Abatacept — Abatacept SC (125 mg) once weekly
  Other Names: BMS-188667; Orencia®
Drug: Adalimumab — Adalimumab SC (40 mg) once every 2 weeks
  Other Names: Humira®
  Arms: Arm 2: (Adalimumab + Methotrexate) followed by (Abatacept + Methotrexate)
Drug: Methotrexate — Methotrexate oral/parenteral maximum tolerated dose (minimum 15 mg and maximum 25 mg weekly)

SUMMARY:
The purpose of this study is to evaluate the superiority in efficacy of abatacept compared with adalimumab, on background methotrexate, in adults with early, seropositive, and shared epitope-positive rheumatoid arthritis and an inadequate methotrexate response.

ELIGIBILITY:
Inclusion Criteria:

* Early rheumatoid arthritis (RA), defined as symptoms of RA that started ≤ 12 months prior to screening and satisfied the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria for the classification of RA at some point during the 12-month period
* Naïve to any targeted (biologic or nonbiologic) disease-modifying antirheumatic drugs (DMARDs), conventional synthetic DMARDs other than methotrexate (MTX), or investigational therapies for RA
* Treated with MTX for at least 12 weeks, with a stable dose of oral or parenteral MTX for at least 4 weeks prior to randomization
* Anti-cyclic citrullinated peptide-2 (Anti-CCP-2) test that is > 3× the upper limit of normal and are positive for rheumatoid factor (RF) according to central lab testing during screening
* At least a Disease Activity Score 28-joint count calculated using C-reactive protein (DAS28-CRP) ≥ 3.2 at screening
* At least 3 tender and at least 3 swollen joints at screening and at randomization

Exclusion Criteria:

* Women who are breastfeeding
* Autoimmune disease other than RA (e.g., psoriasis, systemic lupus erythematosus [SLE], vasculitis, seronegative spondyloarthritis, inflammatory bowel disease, Sjogren's syndrome) or currently active fibromyalgia
* History of or current inflammatory joint disease other than RA (e.g., psoriatic arthritis, gout, reactive arthritis, Lyme disease)
* At risk for tuberculosis
* Recent acute infection
* History of chronic or recurrent bacterial infection (e.g., chronic pyelonephritis, osteomyelitis, bronchiectasis)
* History of infection of a joint prosthesis or artificial joint
* History of systemic fungal infections (such as histoplasmosis, blastomycosis, or coccidiomycosis)
* History of primary immunodeficiency
* Current clinical findings or a history of a demyelinating disorder
* 5 or more joints cannot be assessed for tenderness or swelling

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2027-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (75):
- United States (14):
  - Local Institution - 0036, Fullerton, California
  - Local Institution - 0086, Los Alamitos, California
  - Local Institution - 0041, Aurora, Colorado
  - Local Institution - 0058, Cumberland, Maryland
  - Local Institution - 0038, Hagerstown, Maryland
  - Local Institution - 0084, Eagan, Minnesota
  - Local Institution - 0040, Freehold, New Jersey
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - Local Institution - 0082, Wilmington, North Carolina
  - Local Institution - 0127, Portland, Oregon
  - Local Institution - 0031, Duncansville, Pennsylvania
  - Local Institution - 0034, Jackson, Tennessee
  - Local Institution - 0044, Dallas, Texas
  - Local Institution - 0119, Milwaukee, Wisconsin
- Argentina (8):
  - Local Institution - 0012, CABA, Buenos Aires
  - Local Institution - 0016, Quilmes, Buenos Aires
  - Local Institution - 0014, San Isidro, Buenos Aires
  - Local Institution - 0057, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0022, Buenos Aires
  - Local Institution - 0023, Buenos Aires
  - Local Institution - 0015, Buenos Aires
  - Local Institution - 0099, Córdoba
- Australia (7):
  - Local Institution - 0072, Botany, New South Wales
  - Local Institution - 0062, Paramatta, New South Wales
  - Local Institution - 0063, Maroochydore, Queensland
  - Local Institution - 0102, Woodville South, South Australia
  - Local Institution - 0064, Camberwell, Victoria
  - Local Institution - 0065, Geelong, Victoria
  - Local Institution - 0105, Ivanhoe, Victoria
- Czechia (2):
  - Local Institution - 0028, Brno
  - Local Institution - 0025, Prague
- France (4):
  - Local Institution - 0001, Montpellier
  - Local Institution - 0047, Rouen
  - Local Institution - 0035, Strasbourg
  - Local Institution - 0002, Toulouse
- Germany (5):
  - Local Institution - 0059, Berlin
  - Local Institution - 0055, Bonn
  - Local Institution - 0091, Freiburg im Breisgau
  - Local Institution - 0053, Hamburg
  - Local Institution - 0056, Planegg
- Italy (4):
  - Local Institution - 0083, Catania
  - Local Institution - 0077, Pavia
  - Local Institution - 0078, Perugia
  - Local Institution - 0100, Roma
- Japan (8):
  - Local Institution - 0093, Nagoya, Aichi-ken
  - Local Institution - 0079, Kitakyushu, Fukuoka
  - Local Institution - 0110, Sapporo, Hokkaido
  - Local Institution - 0046, Sendai, Miyagi
  - Local Institution - 0112, Sasebo, Nagasaki
  - Local Institution - 0090, Kawagoe, Saitama
  - Local Institution - 0089, Tokyo
  - Local Institution - 0010, Tokyo
- Mexico (7):
  - Local Institution - 0017, Guadalajara, Jalisco
  - Local Institution - 0117, Guadalajara, Jalisco
  - Local Institution - 0006, Mexico City, Mexico City
  - Local Institution - 0008, Mexico City, Mexico City
  - Local Institution - 0118, San Luis Potosí City, San Luis Potosí
  - Local Institution - 0005, Mérida, Yucatán
  - Local Institution - 0009, Chihuahua City
- Poland (3):
  - Local Institution - 0020, Torun, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0124, Bydgoszcz
  - Local Institution - 0019, Elblag
- Spain (3):
  - Local Institution - 0004, A Coruña
  - Local Institution - 0003, Madrid
  - Local Institution - 0085, Santander
- Switzerland (2):
  - Local Institution - 0049, Basel
  - Local Institution - 0052, Sankt Gallen
- Taiwan (5):
  - Local Institution - 0098, Kaohsiung Niao Sung Dist
  - Local Institution - 0104, New Taipei City
  - Local Institution - 0095, Taichung
  - Local Institution - 0096, Taichung
  - Local Institution - 0120, Tainan
- United Kingdom (3):
  - Local Institution - 0111, Cannock, Staffordshire
  - Local Institution - 0060, Hull
  - Local Institution - 0114, London

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 338 participants were treated during the single-blind treatment. 321 of the participants who completed the single-blind treatment continued to be treated in the open-label.
Groups:
- Abatacept: Participants self-administered Abatacept 125 mg subcutaneous injection weekly up to and including Week 103 (Day 722) with background stable methotrexate therapy
- Adalimumab, Then Abatacept (OLE Period): Participants self-administered Adalimumab 40 mg subcutaneous injection once every 2 weeks up to and including Week 22 (Day 155) with background stable methotrexate therapy. Those participants who entered the OL phase then took 125 mg Abatacept, which was self-administered subcutaneous weekly up to and including Week 103 (Day 722)
Period: Overall Study
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Started (Started=Treated during Single-Blind Treatment) | 169 | 169
Treated in Open-Label (At week 24, all participants ongoing in the OL self-administered abatacept 125 mg subcutaneous weekly up to and including Week 103 (Day 722)) | 160 | 161
Completed (Completed=Completed Single-Blind Treatment) | 162 | 162
Not Completed | 7 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Participant request to discontinue study treatment | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — other reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period) | Total
Number analyzed (Participants) | 169 | 169 | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (13.71) | 47.4 (13.43) | 48.4 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 138 | 268
  Male | 39 | 31 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 9 | 18
  Asian | 17 | 23 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 122 | 113 | 235
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 23 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of SE+ Participants Meeting 50% Improvement in American College of Rheumatology Criteria (ACR50) Response at Week 24
Description: The ACR 50 definition of improvement is a 50% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 50% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication.
Time Frame: Baseline, week 24
Population: All participants that are shared epitope-positive (SE+) at baseline. SE+ participants with missing data at week 24 or discontinuation due to any reason before week 24 are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants | 59.0 [49.5 to 68.0] | 60.3 [50.8 to 69.3]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9026, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.6]

2. Secondary Outcome: Percentage of SE+ Participants Achieving Disease Activity Score 28 Joint Count Calculated Using C Reactive Protein Remission (DAS28-CRP < 2.6) at Week 24
Description: DAS28-CRP is a continuous variable which is a composite of 4 variables: the number of tender joints out of a pre-specified 28 joints, the number of swollen joints out of a pre-specified 28 joints, C-reactive protein in mg/L (CRP) and participant assessment of disease activity measure on a visual analogue scale (VAS) of 100mm. DAS28-CRP scores range from 0 to 10; higher scores indicate more active disease. DAS28-CRP is calculated using the following formula: DAS28-CRP(4) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96 where t28 = number of painful joints from 28 joints, sw28 = number of swollen joints from 28 joints, CRP = c-reactive protein in mg/L, and GH = general health or patient's global assessment of disease activity on a 100 mm VAS.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants | 44.4 [35.3 to 53.9] | 46.6 [37.2 to 56.0]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5824, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.5]

3. Secondary Outcome: Percentage of Participants Meeting 50% Improvement in American College of Rheumatology Criteria (ACR50) Response at Week 24
Description: as for outcome 1
Time Frame: Baseline, week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants | 59.2 [51.4 to 66.7] | 63.9 [56.2 to 71.1]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3534, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI [0.5 to 1.3]

4. Secondary Outcome: Percentage of SE+ Participants Achieving Clinical Disease Activity Index Remission (CDAI <= 2.8) at Week 24
Description: CDAI is a simple linear sum of the following four components: Tender joint counts out of 28 joints, Swollen joint counts out of 28 joints, Participant global assessment of disease activity (0-10cm), Physicians global assessment of disease activity (0-10cm). CDAI scores range from 2-76; higher scores indicate more active disease. CDAI is calculated using the following formula: TJC + SJC + PGA + MDGA where TJC = number of painful joints from 28 joints, SJC = number of swollen joints from 28 joints, PGA = patient global assessment on a visual analog scale 0-10 cm, and MDGA = physician global assessment on a visual analog scale 0-10 cm.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants | 33.3 [24.9 to 42.6] | 35.3 [26.7 to 44.8]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6140, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.5]

5. Secondary Outcome: Adjusted Mean Change From Baseline in SE+ Participant-Reported Pain Visual Analog Scale (VAS) at Week 24
Description: Participant-reported pain by a 0-100mm visual analog scale; higher score indicates more pain. Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline = Post-baseline - Baseline value.
Time Frame: Baseline, week 24
Population: All participants that are shared epitope-positive (SE+) at baseline with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 110 | 107
Score on a scale | -40.9 (2.256) | -37.7 (2.288)

6. Secondary Outcome: Percentage of SE+ Participants Meeting 20% Improvement in American College of Rheumatology Criteria (ACR20) Response Over Time
Description: The ACR 20 definition of improvement is a 20% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 20% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All participants that are shared epitope-positive (SE+) at baseline. SE+ participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 47.0 [37.7 to 56.5] | 51.7 [42.3 to 61.1]
  Day 57 | 66.7 [57.4 to 75.1] | 71.6 [62.4 to 79.5]
  Day 85 | 74.4 [65.5 to 82.0] | 75.9 [67.0 to 83.3]
  Day 113 | 85.5 [77.8 to 91.3] | 76.7 [68.0 to 84.1]
  Day 141 | 82.9 [74.8 to 89.2] | 79.3 [70.8 to 86.3]
  Day 169 | 76.9 [68.2 to 84.2] | 75.9 [67.0 to 83.3]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4996, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4490, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8090, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.7]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.0739, Regression, Logistic; Adjusted Odds Ratio = 1.9, 95% CI 2-sided [0.9 to 3.6]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4201, Regression, Logistic; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.7 to 2.6]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7928, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.6 to 2.0]

7. Secondary Outcome: Percentage of SE+ Participants Meeting 50% Improvement in American College of Rheumatology Criteria (ACR50) Response Over Time
Description: as for outcome 1
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 20.5 [13.6 to 29.0] | 26.7 [18.9 to 35.7]
  Day 57 | 38.5 [29.6 to 47.9] | 43.1 [33.9 to 52.6]
  Day 85 | 54.7 [45.2 to 63.9] | 54.3 [44.8 to 63.6]
  Day 113 | 60.7 [51.2 to 69.6] | 59.5 [50.0 to 68.5]
  Day 141 | 60.7 [51.2 to 69.6] | 60.3 [50.8 to 69.3]
  Day 169 | 59.0 [49.5 to 68.0] | 60.3 [50.8 to 69.3]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.2701, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.4 to 1.3]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4863, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9513, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8536, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.6 to 1.8]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9223, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9026, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.6]

8. Secondary Outcome: Percentage of SE+ Participants Meeting 70% Improvement in American College of Rheumatology Criteria (ACR70) Response Over Time
Description: The ACR 70 definition of improvement is a 70% improvement over baseline in tender and swollen joint counts (#1 and #2) and a 70% improvement in 3 of the 5 remaining core data set measures (Participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, and acute phase reactant value). Baseline value is the last assessment taken prior to first dose of single-blind study medication.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 6.8 [3.0 to 13.0] | 10.3 [5.5 to 17.4]
  Day 57 | 17.9 [11.5 to 26.1] | 24.1 [16.7 to 33.0]
  Day 85 | 30.8 [22.6 to 40.0] | 35.3 [26.7 to 44.8]
  Day 113 | 35.0 [26.5 to 44.4] | 35.3 [26.7 to 44.8]
  Day 141 | 40.2 [31.2 to 49.6] | 44.0 [34.8 to 53.5]
  Day 169 | 39.3 [30.4 to 48.8] | 47.4 [38.1 to 56.9]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3411, Regression, Logistic; Adjusted Odds Ratio = 0.6, 95% CI 2-sided [0.2 to 1.6]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.2546, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.4 to 1.3]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4558, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9544, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5450, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.2227, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.4 to 1.2]

9. Secondary Outcome: Percentage of SE+ Participants Achieving Disease Activity Score 28 Joint Count Calculated Using C Reactive Protein Remission (DAS28-CRP < 2.6) Over Time
Description: as for outcome 2
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 12.8 [7.4 to 20.3] | 16.4 [10.2 to 24.4]
  Day 57 | 30.8 [22.6 to 40.0] | 32.8 [24.3 to 42.1]
  Day 85 | 41.0 [32.0 to 50.5] | 40.5 [31.5 to 50.0]
  Day 113 | 49.6 [40.2 to 59.0] | 52.6 [43.1 to 61.9]
  Day 141 | 54.7 [45.2 to 63.9] | 52.6 [43.1 to 61.9]
  Day 169 | 44.4 [35.3 to 53.9] | 46.6 [37.2 to 56.0]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3200, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.3 to 1.4]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4992, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.5]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8963, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4544, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8985, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.8]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5824, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.5]

10. Secondary Outcome: Percentage of SE+ Participants Achieving Clinical Disease Activity Index Remission (CDAI <= 2.8) Over Time
Description: as for outcome 4
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 9.4 [4.8 to 16.2] | 6.0 [2.5 to 12.0]
  Day 57 | 17.1 [10.8 to 25.2] | 13.8 [8.1 to 21.4]
  Day 85 | 26.5 [18.8 to 35.5] | 19.8 [13.0 to 28.3]
  Day 113 | 29.1 [21.0 to 38.2] | 32.8 [24.3 to 42.1]
  Day 141 | 34.2 [25.7 to 43.5] | 30.2 [22.0 to 39.4]
  Day 169 | 33.3 [24.9 to 42.6] | 35.3 [26.7 to 44.8]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4152, Regression, Logistic; Adjusted Odds Ratio = 1.5, 95% CI 2-sided [0.6 to 4.1]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5917, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.6 to 2.5]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3348, Regression, Logistic; Adjusted Odds Ratio = 1.4, 95% CI 2-sided [0.7 to 2.6]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3959, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.4 to 1.4]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6225, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.7 to 2.0]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6140, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.5]

11. Secondary Outcome: Percentage of SE+ Participants Achieving Simple Disease Activity Index Remission (SDAI <= 3.3) Over Time
Description: SDAI is a simple linear sum of the following five components: Tender joint counts out of 28 joints, Swollen joint counts out of 28 joints, Participant global assessment of disease activity (0-10cm), Physicians global assessment of disease activity (0-10cm), high-sensitivity C-reactive protein (hsCRP mg/dL). SDAI total scores range from 0-86; higher scores indicate more active disease. SDAI is calculated using the following formula: TJC + SJC + PGA + MDGA + CRP where TJC = number of painful joints from 28 joints, SJC = number of swollen joints from 28 joints, PGA = patient global assessment on a visual analog scale 0-10 cm, MDGA = physician global assessment on a visual analog scale 0-10 cm, and CRP = c-reactive protein in mg/dL.
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 117 | 116
Percentage of participants
  Day 29 | 9.4 [4.8 to 16.2] | 7.8 [3.6 to 14.2]
  Day 57 | 17.1 [10.8 to 25.2] | 14.7 [8.8 to 22.4]
  Day 85 | 24.8 [17.3 to 33.6] | 19.8 [13.0 to 28.3]
  Day 113 | 31.6 [23.3 to 40.9] | 31.9 [23.6 to 41.2]
  Day 141 | 35.9 [27.2 to 45.3] | 32.8 [24.3 to 42.1]
  Day 169 | 33.3 [24.9 to 42.6] | 34.5 [25.9 to 43.9]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8084, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.4 to 2.9]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7470, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.5 to 2.3]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5233, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.7 to 2.3]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7295, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.6]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7621, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.6 to 1.9]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6861, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.6]

12. Secondary Outcome: Percentage of Participants Meeting 20% Improvement in American College of Rheumatology Criteria (ACR20) Response Over Time
Description: as for outcome 6
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 46.7 [39.0 to 54.6] | 52.1 [44.3 to 59.8]
  Day 57 | 66.3 [58.6 to 73.4] | 68.6 [61.1 to 75.5]
  Day 85 | 72.8 [65.4 to 79.3] | 76.3 [69.2 to 82.5]
  Day 113 | 85.2 [78.9 to 90.2] | 79.9 [73.0 to 85.6]
  Day 141 | 84.0 [77.6 to 89.2] | 79.9 [73.0 to 85.6]
  Day 169 | 77.5 [70.5 to 83.6] | 76.9 [69.8 to 83.0]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3117, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.2]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6120, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.6 to 1.4]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4339, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.1963, Regression, Logistic; Adjusted Odds Ratio = 1.5, 95% CI 2-sided [0.8 to 2.6]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3275, Regression, Logistic; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.8 to 2.3]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9113, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.7]

13. Secondary Outcome: Percentage of Participants Meeting 50% Improvement in American College of Rheumatology Criteria (ACR50) Response Over Time
Description: as for outcome 1
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 20.1 [14.4 to 27.0] | 27.2 [20.7 to 34.6]
  Day 57 | 38.5 [31.1 to 46.2] | 41.4 [33.9 to 49.2]
  Day 85 | 52.7 [44.9 to 60.4] | 53.3 [45.4 to 61.0]
  Day 113 | 60.4 [52.6 to 67.8] | 59.8 [52.0 to 67.2]
  Day 141 | 61.5 [53.8 to 68.9] | 58.6 [50.8 to 66.1]
  Day 169 | 59.2 [51.4 to 66.7] | 63.9 [56.2 to 71.1]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.1247, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.4 to 1.1]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5656, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.6 to 1.4]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8970, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.5]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9175, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.7 to 1.6]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5996, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3534, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.3]

14. Secondary Outcome: Percentage of Participants Meeting 70% Improvement in American College of Rheumatology Criteria (ACR70) Response Over Time
Description: as for outcome 8
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 5.9 [2.9 to 10.6] | 10.1 [6.0 to 15.6]
  Day 57 | 20.7 [14.9 to 27.6] | 23.1 [17.0 to 30.2]
  Day 85 | 30.2 [23.4 to 37.7] | 32.0 [25.0 to 39.6]
  Day 113 | 35.5 [28.3 to 43.2] | 33.7 [26.6 to 41.4]
  Day 141 | 40.2 [32.8 to 48.0] | 40.8 [33.3 to 48.6]
  Day 169 | 39.1 [31.7 to 46.8] | 45.0 [37.3 to 52.8]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.1641, Regression, Logistic; Adjusted Odds Ratio = 0.6, 95% CI 2-sided [0.2 to 1.3]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5905, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.5]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7146, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.6 to 1.5]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7416, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9026, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.6 to 1.5]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.2605, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.2]

15. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score 28 Joint Count Calculated Using C Reactive Protein Remission (DAS28-CRP < 2.6) Over Time
Description: as for outcome 2
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 10.7 [6.4 to 16.3] | 16.6 [11.3 to 23.0]
  Day 57 | 27.2 [20.7 to 34.6] | 33.7 [26.6 to 41.4]
  Day 85 | 37.3 [30.0 to 45.0] | 40.8 [33.3 to 48.6]
  Day 113 | 49.7 [41.9 to 57.5] | 54.4 [46.6 to 62.1]
  Day 141 | 54.4 [46.6 to 62.1] | 51.5 [43.7 to 59.2]
  Day 169 | 46.7 [39.0 to 54.6] | 50.9 [43.1 to 58.6]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.1078, Regression, Logistic; Adjusted Odds Ratio = 0.6, 95% CI 2-sided [0.3 to 1.1]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.1855, Regression, Logistic; Adjusted Odds Ratio = 0.7, 95% CI 2-sided [0.4 to 1.2]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5223, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.6 to 1.4]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4078, Regression, Logistic; Adjusted Odds Ratio = 0.8, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5238, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4740, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.3]

16. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index Remission (CDAI <= 2.8) Over Time
Description: as for outcome 4
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 7.7 [4.2 to 12.8] | 6.5 [3.3 to 11.3]
  Day 57 | 15.4 [10.3 to 21.7] | 14.2 [9.3 to 20.4]
  Day 85 | 24.9 [18.5 to 32.1] | 20.7 [14.9 to 27.6]
  Day 113 | 31.4 [24.5 to 38.9] | 29.0 [22.3 to 36.5]
  Day 141 | 34.3 [27.2 to 42.0] | 29.0 [22.3 to 36.5]
  Day 169 | 33.7 [26.6 to 41.4] | 32.5 [25.5 to 40.2]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6565, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.5 to 2.9]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7010, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.6 to 2.1]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3683, Regression, Logistic; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.8 to 2.1]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6372, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.2922, Regression, Logistic; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.8178, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.7]

17. Secondary Outcome: Percentage of Participants Achieving Simple Disease Activity Index Remission (SDAI <= 3.3) Over Time
Description: as for outcome 11
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: All treated participants. Participants with missing data at each timepoint are considered non-responders
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 169 | 169
Percentage of participants
  Day 29 | 7.7 [4.2 to 12.8] | 7.7 [4.2 to 12.8]
  Day 57 | 14.8 [9.8 to 21.1] | 16.0 [10.8 to 22.4]
  Day 85 | 23.1 [17.0 to 30.2] | 20.7 [14.9 to 27.6]
  Day 113 | 33.1 [26.1 to 40.8] | 28.4 [21.7 to 35.8]
  Day 141 | 35.5 [28.3 to 43.2] | 28.4 [21.7 to 35.8]
  Day 169 | 34.3 [27.2 to 42.0] | 31.4 [24.5 to 38.9]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.9599, Regression, Logistic; Adjusted Odds Ratio = 1.0, 95% CI 2-sided [0.4 to 2.2]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.7899, Regression, Logistic; Adjusted Odds Ratio = 0.9, 95% CI 2-sided [0.5 to 1.7]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.6305, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.9]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.3491, Regression, Logistic; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.4916, Regression, Logistic; Adjusted Odds Ratio = 1.2, 95% CI 2-sided [0.7 to 1.9]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept vs. Adalimumab; p = 0.5697, Regression, Logistic; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.7 to 1.8]

18. Secondary Outcome: Adjusted Mean Change From Baseline in Disease Activity Score 28 Joint Count Calculated Using C Reactive Protein (DAS28-CRP) Over Time for SE+ Participants
Description: DAS28-CRP is a continuous variable which is a composite of 4 variables: the number of tender joints out of a pre-specified 28 joints, the number of swollen joints out of a pre-specified 28 joints, C-reactive protein in mg/L (CRP) and participant assessment of disease activity measure on a visual analogue scale (VAS) of 100mm. DAS28-CRP scores range from 0 to 10; higher scores indicate more active disease. Remission was defined as DAS28-CRP < 2.6. DAS28-CRP is calculated using the following formula: DAS28-CRP(4) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96 where t28 = number of painful joints from 28 joints, sw28 = number of swollen joints from 28 joints, CRP = c-reactive protein in mg/L, and GH = general health or patient's global assessment of disease activity on a 100 mm VAS. Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline = Post-baseline - Baseline value.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All participants that are shared epitope-positive (SE+) at baseline with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 115 | 113
score on a scale
  Day 29: number analyzed (Participants) | 112 | 113
  Day 29 | -1.3 (0.099) | -1.6 (0.099)
  Day 57: number analyzed (Participants) | 114 | 105
  Day 57 | -2.0 (0.104) | -2.1 (0.109)
  Day 85: number analyzed (Participants) | 112 | 106
  Day 85 | -2.3 (0.109) | -2.4 (0.112)
  Day 113: number analyzed (Participants) | 115 | 111
  Day 113 | -2.7 (0.099) | -2.6 (0.101)
  Day 141: number analyzed (Participants) | 113 | 110
  Day 141 | -2.7 (0.101) | -2.6 (0.102)
  Day 169: number analyzed (Participants) | 109 | 105
  Day 169 | -2.6 (0.114) | -2.6 (0.116)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.0977, longitudinal; Adjusted Mean Difference = 0.2, 95% CI 2-sided [-0.0 to 0.5]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.2889, longitudinal; Adjusted Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.7676, longitudinal; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.6157, longitudinal; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.3904, longitudinal; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.8359, longitudinal; Adjusted Mean Difference = -0.0, 95% CI 2-sided [-0.4 to 0.3]

19. Secondary Outcome: Adjusted Mean Change From Baseline in Clinical Disease Activity Index (CDAI) Over Time for SE+ Participants
Description: CDAI is a simple linear sum of the following four components: Tender joint counts out of 28 joints, Swollen joint counts out of 28 joints, Participant global assessment of disease activity (0-10cm), Physicians global assessment of disease activity (0-10cm). CDAI scores range from 2-76; higher scores indicate more active disease. CDAI remission was defined as =<2.8. CDAI is calculated using the following formula: TJC + SJC + PGA + MDGA where TJC = number of painful joints from 28 joints, SJC = number of swollen joints from 28 joints, PGA = patient global assessment on a visual analog scale 0-10 cm, and MDGA = physician global assessment on a visual analog scale 0-10 cm. Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline = Post-baseline - Baseline value.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 113 | 114
score on a scale
  Day 29: number analyzed (Participants) | 110 | 114
  Day 29 | -15.5 (0.972) | -15.9 (0.955)
  Day 57: number analyzed (Participants) | 113 | 108
  Day 57 | -21.3 (0.928) | -21.9 (0.949)
  Day 85: number analyzed (Participants) | 110 | 106
  Day 85 | -24.6 (0.928) | -23.7 (0.945)
  Day 113: number analyzed (Participants) | 113 | 110
  Day 113 | -26.8 (0.798) | -25.6 (0.808)
  Day 141: number analyzed (Participants) | 108 | 109
  Day 141 | -27.3 (0.783) | -25.6 (0.780)
  Day 169: number analyzed (Participants) | 104 | 104
  Day 169 | -26.9 (0.959) | -25.5 (0.959)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.7852, longitudinal; Adjusted Mean Difference = 0.4, 95% CI 2-sided [-2.3 to 3.1]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.6336, longitudinal; Adjusted Mean Difference = 0.6, 95% CI 2-sided [-2.0 to 3.3]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.4879, longitudinal; Adjusted Mean Difference = -0.9, 95% CI 2-sided [-3.5 to 1.7]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.2812, longitudinal; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-3.5 to 1.0]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.1205, longitudinal; Adjusted Mean Difference = -1.7, 95% CI 2-sided [-3.9 to 0.5]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.3001, longitudinal; Adjusted Mean Difference = -1.4, 95% CI 2-sided [-4.1 to 1.3]

20. Secondary Outcome: Adjusted Mean Change From Baseline in Simple Disease Activity Index (SDAI) Over Time for SE+ Participants
Description: SDAI is a simple linear sum of the following five components: Tender joint counts out of 28 joints, Swollen joint counts out of 28 joints, Participant global assessment of disease activity (0-10cm), Physicians global assessment of disease activity (0-10cm), high-sensitivity C-reactive protein (hsCRP mg/dL). SDAI total scores range from 0-86; higher scores indicate more active disease. Remission was defined as SDAI =< 3.3. SDAI is calculated using the following formula: TJC + SJC + PGA + MDGA + CRP where TJC = number of painful joints from 28 joints, SJC = number of swollen joints from 28 joints, PGA = patient global assessment on a visual analog scale 0-10 cm, MDGA = physician global assessment on a visual analog scale 0-10 cm, and CRP = c-reactive protein in mg/dL. Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline = Post-baseline - Baseline value.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 113 | 113
score on a scale
  Day 29: number analyzed (Participants) | 109 | 113
  Day 29 | -15.6 (1.008) | -16.7 (0.990)
  Day 57: number analyzed (Participants) | 112 | 105
  Day 57 | -21.9 (0.931) | -22.5 (0.962)
  Day 85: number analyzed (Participants) | 109 | 105
  Day 85 | -25.3 (0.935) | -24.6 (0.953)
  Day 113: number analyzed (Participants) | 113 | 110
  Day 113 | -27.5 (0.797) | -26.3 (0.807)
  Day 141: number analyzed (Participants) | 108 | 109
  Day 141 | -28.1 (0.791) | -26.4 (0.787)
  Day 169: number analyzed (Participants) | 104 | 103
  Day 169 | -27.6 (0.978) | -26.1 (0.983)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.4107, longitudinal; Adjusted Mean Difference = 1.2, 95% CI 2-sided [-1.6 to 4.0]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.6824, longitudinal; Adjusted Mean Difference = 0.5, 95% CI 2-sided [-2.1 to 3.2]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.5793, longitudinal; Adjusted Mean Difference = -0.7, 95% CI 2-sided [-3.4 to 1.9]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.2883, longitudinal; Adjusted Mean Difference = -1.5, 95% CI 2-sided [-4.2 to 1.2]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.1285, longitudinal; Adjusted Mean Difference = -1.7, 95% CI 2-sided [-3.9 to 0.5]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.2815, longitudinal; Adjusted Mean Difference = -1.5, 95% CI 2-sided [-4.2 to 1.2]

21. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 3-5 Over Time for SE+ Participants
Description: 1. Tender joint count (standard 68 joint count)
  2. Swollen joint count (standard 66 joint count)
  3. Participant global assessment of pain (a 0-100mm visual analog scale with 100 mm being the worst pain)
  4. Participant global assessment of disease activity (a 0-100mm visual analog scale with 100 mm being the highest disease activity)
  5. Physician global assessment of disease activity (a 0-100mm visual analog scale with 100 mm being the worst case)
  6. Participant assessment of physical function Health Assessment Questionnaire Disability Index (HAQ-DI) (increasing scores for the 8 disability categories indicate increasing level of difficulty). HAQDI is calculated by summing the adjusted categories scores and dividing by the number of categories answered
  7. C-reactive protein (increasing levels indicate increasing level of disease) Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline=Post-baseline - Baseline value.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 115 | 114
score on a scale
  Day 29: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 114 | 114
  Day 29: Participants Global Assess Disease Activity (mm) | -20.0 (2.230) | -21.4 (2.230)
  Day 29: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 111 | 114
  Day 29: Physician Global Assess Disease Activity (mm) | -26.8 (1.896) | -27.1 (1.870)
  Day 29: Participants Assessment of Pain (mm): number analyzed (Participants) | 114 | 113
  Day 29: Participants Assessment of Pain (mm) | -19.5 (2.219) | -23.6 (2.229)
  Day 57: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 115 | 108
  Day 57: Participants Global Assess Disease Activity (mm) | -25.7 (2.205) | -28.4 (2.276)
  Day 57: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 113 | 110
  Day 57: Physician Global Assess Disease Activity (mm) | -37.7 (1.782) | -37.6 (1.806)
  Day 57: Participants Assessment of Pain (mm): number analyzed (Participants) | 114 | 109
  Day 57: Participants Assessment of Pain (mm) | -24.8 (2.305) | -29.1 (2.358)
  Day 85: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 113 | 107
  Day 85: Participants Global Assess Disease Activity (mm) | -33.4 (2.239) | -32.9 (2.302)
  Day 85: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 111 | 109
  Day 85: Physician Global Assess Disease Activity (mm) | -43.8 (1.660) | -42.2 (1.675)
  Day 85: Participants Assessment of Pain (mm): number analyzed (Participants) | 114 | 110
  Day 85: Participants Assessment of Pain (mm) | -33.1 (2.321) | -33.3 (2.363)
  Day 113: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 115 | 111
  Day 113: Participants Global Assess Disease Activity (mm) | -37.7 (2.124) | -35.7 (2.162)
  Day 113: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 113 | 110
  Day 113: Physician Global Assess Disease Activity (mm) | -47.6 (1.462) | -45.8 (1.482)
  Day 113: Participants Assessment of Pain (mm): number analyzed (Participants) | 113 | 110
  Day 113: Participants Assessment of Pain (mm) | -37.0 (2.207) | -34.3 (2.237)
  Day 141: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 113 | 110
  Day 141: Participants Global Assess Disease Activity (mm) | -38.8 (2.243) | -35.0 (2.274)
  Day 141: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 108 | 109
  Day 141: Physician Global Assess Disease Activity (mm) | -48.9 (1.498) | -45.7 (1.491)
  Day 141: Participants Assessment of Pain (mm): number analyzed (Participants) | 111 | 110
  Day 141: Participants Assessment of Pain (mm) | -39.0 (2.212) | -38.3 (2.223)
  Day 169: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 111 | 107
  Day 169: Participants Global Assess Disease Activity (mm) | -39.6 (2.237) | -36.0 (2.278)
  Day 169: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 106 | 106
  Day 169: Physician Global Assess Disease Activity (mm) | -48.0 (1.683) | -45.9 (1.683)
  Day 169: Participants Assessment of Pain (mm): number analyzed (Participants) | 110 | 107
  Day 169: Participants Assessment of Pain (mm) | -40.9 (2.256) | -37.7 (2.288)

22. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 1-2 Over Time for SE+ Participants
Description: as for outcome 21
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: Joints count
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 115 | 114
Joints count
  Day 29: Total Tender Joint Count: number analyzed (Participants) | 114 | 114
  Day 29: Total Tender Joint Count | -9.1 (0.580) | -8.6 (0.580)
  Day 29: Total Swollen Joint Count: number analyzed (Participants) | 114 | 114
  Day 29: Total Swollen Joint Count | -6.2 (0.422) | -6.7 (0.422)
  Day 57: Total Tender Joint Count: number analyzed (Participants) | 115 | 110
  Day 57: Total Tender Joint Count | -11.9 (0.608) | -11.6 (0.621)
  Day 57: Total Swollen Joint Count: number analyzed (Participants) | 115 | 110
  Day 57: Total Swollen Joint Count | -8.6 (0.378) | -8.8 (0.386)
  Day 85: Total Tender Joint Count: number analyzed (Participants) | 114 | 110
  Day 85: Total Tender Joint Count | -13.5 (0.608) | -12.7 (0.618)
  Day 85: Total Swollen Joint Count: number analyzed (Participants) | 114 | 110
  Day 85: Total Swollen Joint Count | -9.5 (0.352) | -9.4 (0.358)
  Day 113: Total Tender Joint Count: number analyzed (Participants) | 115 | 111
  Day 113: Total Tender Joint Count | -14.5 (0.516) | -13.8 (0.526)
  Day 113: Total Swollen Joint Count: number analyzed (Participants) | 115 | 111
  Day 113: Total Swollen Joint Count | -10.1 (0.321) | -9.8 (0.326)
  Day 141: Total Tender Joint Count: number analyzed (Participants) | 113 | 110
  Day 141: Total Tender Joint Count | -14.8 (0.499) | -13.9 (0.506)
  Day 141: Total Swollen Joint Count: number analyzed (Participants) | 113 | 110
  Day 141: Total Swollen Joint Count | -10.4 (0.321) | -9.8 (0.325)
  Day 169: Total Tender Joint Count: number analyzed (Participants) | 109 | 108
  Day 169: Total Tender Joint Count | -14.7 (0.580) | -13.8 (0.583)
  Day 169: Total Swollen Joint Count: number analyzed (Participants) | 109 | 108
  Day 169: Total Swollen Joint Count | -10.2 (0.397) | -9.7 (0.399)

23. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 6 Over Time for SE+ Participants
Description: 6) Participant assessment of physical function Health Assessment Questionnaire Disability Index (HAQ-DI). For the eight disability categories (Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities), there is an aids or devices variables to record the type of assistance. If aids or devices and/or assistance from another person are checked for a category, the score is set to 2 (much difficulty), if the original score is 0 (no difficulty) or 1 (some difficulty). HAQ-DI is then calculated by summing the adjusted categories scores and dividing by the number of categories answered (increasing scores for the 8 disability categories questionnaire indicate increasing level of difficulty with 0 being the lowest score "without any difficulty" and 3 being the highest score "unable to do".
  Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline=Post-baseline - Baseline value.
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 115 | 114
score on a scale
  Day 29: Disability Index: number analyzed (Participants) | 114 | 114
  Day 29: Disability Index | -0.4 (0.047) | -0.5 (0.047)
  Day 57: Disability Index: number analyzed (Participants) | 115 | 109
  Day 57: Disability Index | -0.6 (0.049) | -0.6 (0.050)
  Day 85: Disability Index: number analyzed (Participants) | 113 | 109
  Day 85: Disability Index | -0.8 (0.050) | -0.7 (0.051)
  Day 113: Disability Index: number analyzed (Participants) | 114 | 110
  Day 113: Disability Index | -0.8 (0.047) | -0.7 (0.048)
  Day 141: Disability Index: number analyzed (Participants) | 110 | 110
  Day 141: Disability Index | -0.9 (0.046) | -0.8 (0.046)
  Day 169: Disability Index: number analyzed (Participants) | 110 | 108
  Day 169: Disability Index | -0.9 (0.049) | -0.8 (0.050)

24. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 7 Over Time for SE+ Participants
Description: as for outcome 21
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: as for outcome 18
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 115 | 114
mg/L
  Day 29: C Reactive Protein (mg/L): number analyzed (Participants) | 114 | 114
  Day 29: C Reactive Protein (mg/L) | -1.4 (1.986) | -8.1 (1.995)
  Day 57: C Reactive Protein (mg/L): number analyzed (Participants) | 114 | 107
  Day 57: C Reactive Protein (mg/L) | -6.1 (0.818) | -7.4 (0.845)
  Day 85: C Reactive Protein (mg/L): number analyzed (Participants) | 113 | 109
  Day 85: C Reactive Protein (mg/L) | -6.7 (0.745) | -8.6 (0.759)
  Day 113: C Reactive Protein (mg/L): number analyzed (Participants) | 115 | 111
  Day 113: C Reactive Protein (mg/L) | -7.5 (0.701) | -7.3 (0.713)
  Day 141: C Reactive Protein (mg/L): number analyzed (Participants) | 113 | 110
  Day 141: C Reactive Protein (mg/L) | -7.9 (0.724) | -7.6 (0.733)
  Day 169: C Reactive Protein (mg/L): number analyzed (Participants) | 111 | 108
  Day 169: C Reactive Protein (mg/L) | -6.6 (1.083) | -5.4 (1.098)

25. Secondary Outcome: Adjusted Mean Change From Baseline in Disease Activity Score 28 Joint Count Calculated Using C Reactive Protein (DAS28-CRP) Over Time for All Participants
Description: as for outcome 18
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 165 | 164
score on a scale
  Day 29: number analyzed (Participants) | 164 | 164
  Day 29 | -1.2 (0.084) | -1.5 (0.084)
  Day 57: number analyzed (Participants) | 163 | 158
  Day 57 | -1.9 (0.089) | -2.1 (0.089)
  Day 85: number analyzed (Participants) | 163 | 158
  Day 85 | -2.2 (0.091) | -2.4 (0.091)
  Day 113: number analyzed (Participants) | 165 | 163
  Day 113 | -2.6 (0.084) | -2.6 (0.084)
  Day 141: number analyzed (Participants) | 163 | 161
  Day 141 | -2.7 (0.085) | -2.5 (0.085)
  Day 169: number analyzed (Participants) | 157 | 157
  Day 169 | -2.6 (0.094) | -2.6 (0.093)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.0099, longitudinal; Adjusted Mean Difference = 0.3, 95% CI 2-sided [0.1 to 0.5]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.1519, longitudinal; Adjusted Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.2505, longitudinal; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.5248, longitudinal; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.1778, longitudinal; Adjusted Mean Difference = -0.0, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.8510, longitudinal; Adjusted Mean Difference = -0.0, 95% CI 2-sided [-0.3 to 0.2]

26. Secondary Outcome: Adjusted Mean Change From Baseline in Clinical Disease Activity Index (CDAI) Over Time for All Participants
Description: as for outcome 19
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 163 | 163
score on a scale
  Day 29: number analyzed (Participants) | 162 | 163
  Day 29 | -14.6 (0.818) | -15.9 (0.823)
  Day 57: number analyzed (Participants) | 162 | 160
  Day 57 | -20.9 (0.786) | -21.6 (0.784)
  Day 85: number analyzed (Participants) | 161 | 157
  Day 85 | -23.5 (0.763) | -23.5 (0.769)
  Day 113: number analyzed (Participants) | 163 | 161
  Day 113 | -26.6 (0.644) | -25.4 (0.646)
  Day 141: number analyzed (Participants) | 155 | 161
  Day 141 | -27.1 (0.647) | -25.2 (0.631)
  Day 169: number analyzed (Participants) | 152 | 156
  Day 169 | -26.7 (0.763) | -25.4 (0.749)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.2319, longitudinal; Adjusted Mean Difference = 1.3, 95% CI 2-sided [-0.9 to 3.5]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.5572, longitudinal; Adjusted Mean Difference = 0.6, 95% CI 2-sided [-1.5 to 2.7]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.9366, longitudinal; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-2.0 to 2.1]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.1508, longitudinal; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-3.5 to 1.0]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.0303, longitudinal; Adjusted Mean Difference = -1.9, 95% CI 2-sided [-3.6 to -0.2]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.2333, longitudinal; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-3.3 to 0.8]

27. Secondary Outcome: Adjusted Mean Change From Baseline in Simple Disease Activity Index (SDAI) Over Time for All Participants
Description: as for outcome 20
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 163 | 162
Score on a scale
  Day 29: number analyzed (Participants) | 161 | 162
  Day 29 | -14.7 (0.843) | -16.6 (0.849)
  Day 57: number analyzed (Participants) | 161 | 157
  Day 57 | -21.5 (0.788) | -22.1 (0.789)
  Day 85: number analyzed (Participants) | 160 | 156
  Day 85 | -24.0 (0.769) | -24.2 (0.775)
  Day 113: number analyzed (Participants) | 163 | 161
  Day 113 | -27.2 (0.648) | -26.0 (0.649)
  Day 141: number analyzed (Participants) | 155 | 160
  Day 141 | -27.7 (0.661) | -25.8 (0.647)
  Day 169: number analyzed (Participants) | 151 | 155
  Day 169 | -27.3 (0.787) | -26.0 (0.771)
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 29; Test type: Superiority — Abatacept - Adalimumab; p = 0.0938, longitudinal; Adjusted Mean Difference = 1.9, 95% CI 2-sided [-0.3 to 4.2]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 57; Test type: Superiority — Abatacept - Adalimumab; p = 0.6053, longitudinal; Adjusted Mean Difference = 0.6, 95% CI 2-sided [-1.6 to 2.7]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 85; Test type: Superiority — Abatacept - Adalimumab; p = 0.8570, longitudinal; Adjusted Mean Difference = 0.2, 95% CI 2-sided [-1.9 to 2.3]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 113; Test type: Superiority — Abatacept - Adalimumab; p = 0.1592, longitudinal; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-3.0 to 0.5]
Statistical Analysis 5: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 141; Test type: Superiority — Abatacept - Adalimumab; p = 0.0319, longitudinal; Adjusted Mean Difference = -1.9, 95% CI 2-sided [-3.7 to -0.2]
Statistical Analysis 6: Comparison: Abatacept vs Adalimumab, Then Abatacept (OLE Period); Day 169; Test type: Superiority — Abatacept - Adalimumab; p = 0.2059, longitudinal; Adjusted Mean Difference = -1.3, 95% CI 2-sided [-3.4 to 0.7]

28. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 3-5 Over Time for All Participants
Description: as for outcome 21
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 166 | 166
score on a scale
  Day 29: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 166 | 165
  Day 29: Participants Global Assess Disease Activity (mm) | -19.4 (1.865) | -20.6 (1.868)
  Day 29: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 163 | 165
  Day 29: Physician Global Assess Disease Activity (mm) | -24.4 (1.613) | -27.7 (1.612)
  Day 29: Participants Assessment of Pain (mm) | -19.2 (1.872) | -22.7 (1.863)
  Day 57: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 166 | 161
  Day 57: Participants Global Assess Disease Activity (mm) | -27.3 (1.888) | -28.3 (1.893)
  Day 57: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 163 | 162
  Day 57: Physician Global Assess Disease Activity (mm) | -35.7 (1.583) | -36.7 (1.579)
  Day 57: Participants Assessment of Pain (mm): number analyzed (Participants) | 165 | 162
  Day 57: Participants Assessment of Pain (mm) | -25.9 (1.957) | -28.7 (1.954)
  Day 85: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 164 | 159
  Day 85: Participants Global Assess Disease Activity (mm) | -32.8 (1.874) | -32.8 (1.884)
  Day 85: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 162 | 161
  Day 85: Physician Global Assess Disease Activity (mm) | -40.1 (1.459) | -41.2 (1.459)
  Day 85: Participants Assessment of Pain (mm): number analyzed (Participants) | 164 | 163
  Day 85: Participants Assessment of Pain (mm) | -32.1 (1.939) | -33.7 (1.923)
  Day 113: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 165 | 163
  Day 113: Participants Global Assess Disease Activity (mm) | -37.7 (1.787) | -34.8 (1.780)
  Day 113: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 163 | 161
  Day 113: Physician Global Assess Disease Activity (mm) | -46.8 (1.216) | -44.9 (1.218)
  Day 113: Participants Assessment of Pain (mm): number analyzed (Participants) | 163 | 162
  Day 113: Participants Assessment of Pain (mm) | -36.6 (1.883) | -33.9 (1.871)
  Day 141: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 163 | 162
  Day 141: Participants Global Assess Disease Activity (mm) | -38.4 (1.866) | -34.1 (1.856)
  Day 141: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 155 | 162
  Day 141: Physician Global Assess Disease Activity (mm) | -48.5 (1.258) | -45.2 (1.221)
  Day 141: Participants Assessment of Pain (mm): number analyzed (Participants) | 161 | 163
  Day 141: Participants Assessment of Pain (mm) | -38.7 (1.858) | -35.4 (1.830)
  Day 169: Participants Global Assess Disease Activity (mm): number analyzed (Participants) | 160 | 159
  Day 169: Participants Global Assess Disease Activity (mm) | -39.1 (1.842) | -36.6 (1.827)
  Day 169: Physician Global Assess Disease Activity (mm): number analyzed (Participants) | 154 | 158
  Day 169: Physician Global Assess Disease Activity (mm) | -47.7 (1.320) | -46.2 (1.296)
  Day 169: Participants Assessment of Pain (mm): number analyzed (Participants) | 158 | 159
  Day 169: Participants Assessment of Pain (mm) | -39.5 (1.895) | -37.0 (1.864)

29. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 1-2 Over Time for All Participants
Description: as for outcome 21
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: Joints count
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 166 | 167
Joints count
  Day 29: Total Tender Joint Count | -8.1 (0.529) | -8.2 (0.527)
  Day 29: Total Swollen Joint Count | -6.1 (0.374) | -6.6 (0.372)
  Day 57: Total Tender Joint Count: number analyzed (Participants) | 164 | 163
  Day 57: Total Tender Joint Count | -11.3 (0.549) | -11.1 (0.545)
  Day 57: Total Swollen Joint Count: number analyzed (Participants) | 164 | 163
  Day 57: Total Swollen Joint Count | -8.7 (0.322) | -8.7 (0.319)
  Day 85: Total Tender Joint Count: number analyzed (Participants) | 165 | 163
  Day 85: Total Tender Joint Count | -12.7 (0.507) | -12.4 (0.506)
  Day 85: Total Swollen Joint Count: number analyzed (Participants) | 165 | 163
  Day 85: Total Swollen Joint Count | -9.3 (0.289) | -9.4 (0.289)
  Day 113: Total Tender Joint Count: number analyzed (Participants) | 165 | 163
  Day 113: Total Tender Joint Count | -14.4 (0.411) | -13.9 (0.410)
  Day 113: Total Swollen Joint Count: number analyzed (Participants) | 165 | 163
  Day 113: Total Swollen Joint Count | -10.1 (0.255) | -9.8 (0.254)
  Day 141: Total Tender Joint Count: number analyzed (Participants) | 163 | 163
  Day 141: Total Tender Joint Count | -14.8 (0.417) | -13.8 (0.414)
  Day 141: Total Swollen Joint Count: number analyzed (Participants) | 163 | 163
  Day 141: Total Swollen Joint Count | -10.6 (0.259) | -9.9 (0.257)
  Day 169: Total Tender Joint Count: number analyzed (Participants) | 158 | 160
  Day 169: Total Tender Joint Count | -14.5 (0.474) | -13.8 (0.468)
  Day 169: Total Swollen Joint Count: number analyzed (Participants) | 158 | 160
  Day 169: Total Swollen Joint Count | -10.2 (0.311) | -9.8 (0.307)

30. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 6 Over Time for All Participants
Description: as for outcome 23
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 166 | 165
score on a scale
  Day 29: Disability Index | -0.4 (0.040) | -0.5 (0.040)
  Day 57: Disability Index: number analyzed (Participants) | 166 | 161
  Day 57: Disability Index | -0.6 (0.042) | -0.6 (0.042)
  Day 85: Disability Index: number analyzed (Participants) | 164 | 161
  Day 85: Disability Index | -0.7 (0.043) | -0.6 (0.043)
  Day 113: Disability Index: number analyzed (Participants) | 163 | 161
  Day 113: Disability Index | -0.7 (0.041) | -0.7 (0.041)
  Day 141: Disability Index: number analyzed (Participants) | 160 | 162
  Day 141: Disability Index | -0.8 (0.040) | -0.7 (0.040)
  Day 169: Disability Index: number analyzed (Participants) | 159 | 160
  Day 169: Disability Index | -0.8 (0.042) | -0.8 (0.042)

31. Secondary Outcome: Adjusted Mean Change From Baseline in American College of Rheumatology (ACR) Core Components 7 Over Time for All Participants
Description: as for outcome 21
Time Frame: Baseline, day 29, 57, 85, 113, 141, 169
Population: All treated participants with both baseline and post-baseline measurements. Non-responders are not included
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 166 | 166
mg/L
  Day 29: C Reactive Protein (mg/L) | -1.4 (1.520) | -6.8 (1.514)
  Day 57: C Reactive Protein (mg/L): number analyzed (Participants) | 164 | 160
  Day 57: C Reactive Protein (mg/L) | -5.7 (0.635) | -6.4 (0.635)
  Day 85: C Reactive Protein (mg/L): number analyzed (Participants) | 164 | 162
  Day 85: C Reactive Protein (mg/L) | -5.4 (0.719) | -6.6 (0.717)
  Day 113: C Reactive Protein (mg/L): number analyzed (Participants) | 165 | 163
  Day 113: C Reactive Protein (mg/L) | -5.7 (0.704) | -5.8 (0.702)
  Day 141: C Reactive Protein (mg/L): number analyzed (Participants) | 163 | 162
  Day 141: C Reactive Protein (mg/L) | -5.9 (0.778) | -5.5 (0.774)
  Day 169: C Reactive Protein (mg/L): number analyzed (Participants) | 159 | 160
  Day 169: C Reactive Protein (mg/L) | -6.2 (0.912) | -5.0 (0.900)

32. Secondary Outcome: Adjusted Mean Change From Baseline in 36-item Short Form Survey (SF-36) Over Time for SE+ Participants
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life, which covers 8 health dimensions within 2 components. The physical component summary (PCS) consists of these 4 subscales: Physical functioning, Role-physical, Bodily pain, General health. The mental component summary (MCS) consists of these 4 subscales: Vitality, Social functioning, Role-emotional, Mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100, with a higher score indicating better quality of life. The 8 subscales will be scored using norm-based methods that have standardized the T-scores to a mean of 50 and a standard deviation of 10 in the general population.
Time Frame: Up to week 24
Population: All participants that are shared epitope-positive (SE+) at baseline with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 110 | 109
T-score
  Day 169: Physical Functioning | 9.2 (0.813) | 9.8 (0.817)
  Day 169: Role-Physical: number analyzed (Participants) | 108 | 109
  Day 169: Role-Physical | 9.1 (0.809) | 8.9 (0.805)
  Day 169: Bodily Pain: number analyzed (Participants) | 108 | 109
  Day 169: Bodily Pain | 14.2 (0.863) | 12.0 (0.859)
  Day 169: General Health | 8.1 (0.779) | 6.5 (0.783)
  Day 169: Vitality: number analyzed (Participants) | 108 | 109
  Day 169: Vitality | 10.0 (0.878) | 8.4 (0.874)
  Day 169: Social Functioning: number analyzed (Participants) | 108 | 109
  Day 169: Social Functioning | 9.6 (0.828) | 9.4 (0.824)
  Day 169: Role-Emotional: number analyzed (Participants) | 108 | 109
  Day 169: Role-Emotional | 9.0 (0.921) | 9.1 (0.917)
  Day 169: Mental Health: number analyzed (Participants) | 108 | 109
  Day 169: Mental Health | 8.9 (0.799) | 7.1 (0.795)
  Day 169: Physical Component Summary: number analyzed (Participants) | 108 | 109
  Day 169: Physical Component Summary | 10.2 (0.738) | 9.6 (0.735)
  Day 169: Mental Component Summary: number analyzed (Participants) | 108 | 109
  Day 169: Mental Component Summary | 8.4 (0.818) | 7.3 (0.814)

33. Secondary Outcome: Adjusted Mean Change From Baseline in SF-36 Over Time for All Participants
Description: as for outcome 32
Time Frame: Up to week 24
Population: All treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Abatacept | Adalimumab, Then Abatacept (OLE Period)
Number analyzed (Participants) | 159 | 161
T-score
  Day 169: Physical Functioning | 8.9 (0.706) | 9.4 (0.697)
  Day 169: Role-Physical: number analyzed (Participants) | 157 | 161
  Day 169: Role-Physical | 8.6 (0.681) | 8.7 (0.669)
  Day 169: Bodily Pain: number analyzed (Participants) | 157 | 161
  Day 169: Bodily Pain | 13.5 (0.719) | 11.7 (0.706)
  Day 169: General Health | 7.9 (0.652) | 6.7 (0.644)
  Day 169: Vitality: number analyzed (Participants) | 157 | 161
  Day 169: Vitality | 9.4 (0.740) | 8.8 (0.725)
  Day 169: Social Functioning: number analyzed (Participants) | 157 | 161
  Day 169: Social Functioning | 8.9 (0.701) | 9.8 (0.690)
  Day 169: Role-Emotional: number analyzed (Participants) | 157 | 161
  Day 169: Role-Emotional | 8.4 (0.773) | 8.8 (0.759)
  Day 169: Mental Health: number analyzed (Participants) | 157 | 161
  Day 169: Mental Health | 8.0 (0.712) | 7.6 (0.700)
  Day 169: Physical Component Summary: number analyzed (Participants) | 157 | 161
  Day 169: Physical Component Summary | 9.9 (0.619) | 9.2 (0.608)
  Day 169: Mental Component Summary: number analyzed (Participants) | 157 | 161
  Day 169: Mental Component Summary | 7.6 (0.718) | 7.7 (0.705)

34. Secondary Outcome: Adjusted Mean Change From Baseline in 36-item Short Form Survey (SF-36) at Week 104 for SE+ Participants
Description: The SF-36 v2.0, which covers 8 health dimensions within 2 components. The physical component summary (PCS) of the SF-36 consists of these 4 subscales: Physical functioning, Role-physical, Bodily pain, General health. The mental component summary (MCS) of the SF-36 consists of these 4 subscales: Vitality, Social functioning, Role-emotional, Mental health. The scores range from 0 to 100, with a higher score indicating better quality of life. The 2 summary scores (PCS and MCS) will be calculated by taking a weighted linear combination of the 8 individual subscales. Baseline value is the last assessment taken prior to first dose of single-blind study medication. Change from Baseline = Post-baseline - Baseline value.
Time Frame: Up to week 24
Reporting Status: Not Posted, anticipated posting 2025-12

35. Secondary Outcome: Adjusted Mean Change From Baseline in 36-item Short Form Survey (SF-36) at Week 104 for All Participants
Description: as for outcome 34
Time Frame: Up to week 24
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from first dose till death (Up to 20 months). Serious adverse events and non-serious adverse events were collected from first dose until 56 days after last dose of study therapy (Up to approximately 9 months).
Description: Data at cut-off is only for the single blind treatment period and is prior to the open label extension phase,
Groups:
- Abatacept Only: Participants self-administered Abatacept 125 mg subcutaneous injection weekly up to and including Week 103 (Day 722) with background stable methotrexate therapy
Arm/Group | Abatacept Only | Adalimumab, Then Abatacept (OLE Period)
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/169
Serious Adverse Events (participants affected / at risk) | 4/169 | 6/169
Other Adverse Events (participants affected / at risk) | 34/169 | 41/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Only (N=169) | Adalimumab, Then Abatacept (OLE Period) (N=169)
Atypical pneumonia (Infections and infestations) | 0 | 1
Pilonidal disease (Infections and infestations) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Only (N=169) | Adalimumab, Then Abatacept (OLE Period) (N=169)
COVID-19 (Infections and infestations) | 20 | 23
Nasopharyngitis (Infections and infestations) | 11 | 10
Upper respiratory tract infection (Infections and infestations) | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT04909801/Prot_SAP_000.pdf